CLINICAL TRIAL: NCT02060552
Title: Diacerein Combined With Febuxostat Relieves Symptoms of Gout by Suppressing IL-1βinflammation
Brief Title: Immune Molecular and Inflammatory Cytokines Dysfunction Analysis in Gout Patients With Different Urate Levels
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Yikai Yu, Doctor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Diagout1
Record Dates: First submitted 2014-02-08; First posted 2014-02-12 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Primary Gout
MeSH Terms: interventions — diacerein; Colchicine; Febuxostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Febuxostat (Placebo Comparator): Febuxostat 40mg once a day
  Interventions: Drug: Febuxostat
- Febuxostat plus diacerein (Experimental): Febuxostat 40mg once a day plus diacerein 50mg twice a day
  Interventions: Drug: Diacerein; Drug: Febuxostat
- Febuxostat plus Colchicine (Experimental): Febuxostat 40mg once a day plus Colchicine 0.5mg twice a day
  Interventions: Drug: Colchicine; Drug: Febuxostat

INTERVENTIONS:
Drug: Diacerein — oral administration of IL-1βinhibitory
  Other Names: Diacetylrhein
  Arms: Febuxostat plus diacerein
Drug: Colchicine — Colchicine is a toxic natural product and secondary metabolite, originally extracted from plants of the genus Colchicum (autumn crocus, Colchicum autumnale, also known as "meadow saffron"). It was used originally to treat rheumatic complaints, especially gout as the positive control
  Other Names: Colcrys; Generics
  Arms: Febuxostat plus Colchicine
Drug: Febuxostat — A urate lowering drug, an inhibitor of xanthine oxidase that is indicated for use in the treatment of hyperuricemia and gout
  Other Names: No other names

SUMMARY:
The aim of study was to assess the efficiency and safety of oral IL-1βinhibitor in combination with urate lowering therapy on joint pain intensity,urate control, global assessments of disease activity, self-monitored gouty acute flare times, inflammatory markers and symptoms improving related life quantity in gouty patients.

DETAILED DESCRIPTION:
This was a randomized single-dose, open-label and active-controlled study which was carried out in 96 primary gout patients. Subjects and doctors have no access to randomization sequence which is determined by the primary investigator.All patients received an open-label febuxostat 40mg daily during the whole study. Healthy control were 32 age-matched men from volunteers in the medical health center.Two primary end points included pain intensity measurement which was recorded at each visit and subsequently acute flare times which was recorded at home and reported to investigator.

ELIGIBILITY:
Inclusion Criteria:

All participants who were allocated to the study all had a history of taking tolerable and adequate dose of urate lowering therapy including febuxostat 40-80mg daily or allopurinol 200-300 mg daily for at least 4 weeks and were defined as difficult to treat or refractory gout patients. All patients had a negative of rheumatoid factor and antinuclear antibody, Hb>100g/L, total leukocyte count≥3.5×109, PLT≥80×109, serum creatinine<133umol/L, transaminases<60U/L and fasting urate≥6.0mg/dL.

Inclusion criteria for the gouty patients were age≥18 years old, BMI(18-30kg/m2). All participants enrolled in our study fulfilled American College of Rheumatology criteria for primary gout.

Exclusion Criteria:

Exclusion criteria included secondary gout (because it is always associated with some underlying renal disease), a history of congestive heart failure, serum creatinine≥133umol/L (because the patients have underlying risks if NSAID needed) or the use of glucocorticoid>15mg daily,colchicine, uricosuric drugs, chemotherapy or immunosuppressive therapy in the past three months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Patients'intensity of pain | 12 weeks
  Patients' intensity of pain was assessed at each visit by a single question using a 100mm visual analogue scale (VAS). The pain question was how much pains have you had because of your illness in the past seven days? The two anchors were no pain (0 score) and unbearable pain (score of 100). Patients were instructed to draw a vertical mark on the scaleline and the investigator measured the length and recorded the result.
Acute gout flare times | 24 weeks
  Acute gout flare was defined by pain, redness, swelling, and warmth on joints or adjacent soft tissue and pain VAS more than 3.0. For subsequent gout flares, subjects were recorded events by themselves and were reported to investigator whether they had any new or recurrent gout flares since their last visit

SECONDARY OUTCOMES:
Serum and urine urate concentration | 24 weeks
  serum urate concentration and 24h urine urate concentration
HAQ | 12 weeks
  Healthy Assessment Questionnaire (HAQ) disability index might be valuable to assess the joints function impaired by gout flares.HAQ comprised twenty questions and each question has a corresponding mark : 0, 1 or 2. Sum of each answer of the questions was divided by 20
Flow Cytometry analysis on cell markers | 12 weeks
  Inhibitory T cell:CD4 Help T cell:CD8 Natural Killer cell:CD56,CD69，CD16 and CD25 (CD 56 dim and CD56 bright) B cell:CD19 and CD20
Quantitative PCR for mRNA expression of inflammatory cytokines on PBMC | 12 weeks
  IL-1β,IL-18, IL-10
Serum concentration of inflammatory cytokines | 12 weeks
  IL-1β，IL-10，IL-6 and IL-8 etc.

CONTACTS AND LOCATIONS:
Overall Officials: Shaoxian HU, Doctor, Principal Investigator — Tongji Hospital
Locations (1):
- Yikai YU, Wuhan, Hubei, China